CLINICAL TRIAL: NCT02256475
Title: A Phase 1b, Open-Label, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NBI-98854 in Children and Adolescents With Tourette Syndrome
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of NBI-98854 in Children and Adolescents With Tourette Syndrome
Acronym: T-FORCE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NBI-98854-1403
Record Dates: First submitted 2014-09-23; First posted 2014-10-03 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Adolescents Dose Group 1 (Experimental): Fixed dose of NBI-98854 administered once daily at 0800 for 14 days.
  Interventions: Drug: NBI-98854
- Adolescents Dose Group 2 (Experimental): Fixed dose of NBI-98854 administered once daily at 0800 for 14 days. Dosing will not commence until all safety and PK results from the adolescent dose group 1 have been reviewed to ensure there are no safety concerns and that maximum tolerated dose (MTD) has not been reached.
  Interventions: Drug: NBI-98854
- Adolescents Dose Group 3 (Experimental): Fixed dose of NBI-98854 administered once daily at 0800 for 14 days. Dosing will not commence until all safety and PK results from the adolescent dose group 2 have been reviewed to ensure there are no safety concerns and that MTD has not been reached.
  Interventions: Drug: NBI-98854
- Children Dose Group 1 (Experimental): Fixed dose of NBI-98854 administered once daily at 0800 for 14 days. Dosing will not commence until all safety and PK results from the adolescent dose group 1 have been reviewed to ensure there are no safety concerns and that MTD has not been reached.
  Interventions: Drug: NBI-98854
- Children Dose Group 2 (Experimental): Fixed dose of NBI-98854 administered once daily at 0800 for 14 days. Dosing will not commence until all safety and PK results from the children dose group 1 have been reviewed to ensure there are no safety concerns and that MTD has not been reached.
  Interventions: Drug: NBI-98854
- Children Dose Group 3 (Experimental): Fixed dose of NBI-98854 administered once daily at 0800 for 14 days. Dosing will not commence until all safety and PK results from the children dose group 2 have been reviewed to ensure there are no safety concerns and that MTD has not been reached.
  Interventions: Drug: NBI-98854

INTERVENTIONS:
Drug: NBI-98854

SUMMARY:
This is a Phase 1b, open-label, multiple-dose study of the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of NBI-98854 in a total of 36 pediatric subjects with Tourette syndrome (TS). The study will be conducted in approximately 18 male and female children (6 to 11 years of age) and approximately 18 male and female adolescents (12 to 18 years of age). Both age groups will be divided equally into 3 dosing cohorts with 6 subjects each. Ascending doses will be evaluated as part of a staggered-cohort design. Study drug will be administered in each cohort for 14 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Have documentation of written informed consent, or written and witnessed assent from the subject and written informed consent from the subject's parent or legal guardian.
2. Be in good general health.
3. Have a Diagnostic and Statistical Manual of Mental Disorders diagnosis of Tourette Syndrome (DSM-IV or -V).
4. Have TS symptoms that impair school, occupational, and/or social function.
5. If medications are being used to treat TS symptoms, must be on stable doses of these medications for a minimum of 30 days before baseline (Day -1), and the medication regimen is expected to remain stable throughout the study period. The use of tetrabenazine to treat TS symptoms is prohibited.
6. Subjects of childbearing potential who do not practice total abstinence must be instructed on the proper use of barrier methods of contraception and agree to use hormonal or two forms of nonhormonal contraception consistently from screening until 30 days after the last dose of study drug.
7. Adolescent subjects (12 to 18 years of age) must have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids. Subjects who are on stable doses of prescribed benzodiazepines, opiates, or psychostimulants are allowed to participate in the study.
8. Adolescent subjects (12 to 18 years of age) must have a negative alcohol breath test.
9. Be willing and able to adhere to the study regimen and study procedures described in the protocol and informed consent/assent forms, including all requirements at the study center and return for the follow-up visit.

Exclusion Criteria:

1. Have an unstable medical condition or chronic disease.
2. Had a medically significant illness within 30 days of screening.
3. Excessive use of tobacco and/or nicotine-containing products.
4. Have a history of substance (drug) dependence or substance or alcohol abuse.
5. Are currently pregnant or lactating.
6. Have a known history of neuroleptic malignant syndrome.
7. Have a known history of long QT syndrome or cardiac tachy-arrhythmia.
8. Have a cancer diagnosis within 3 years prior to screening, with the exception of localized skin cancer or carcinoma in situ of the cervix.
9. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
10. Have a significant risk of suicidal or violent behavior.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events following dosing with NBI-98854 | Up to 21 days
Area Under Curve (AUC) of NBI-98854 and its metabolites following repeated daily doses of NBI-98854 | Day 1: predose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose; Day 14: predose, 0.5, 1, 2, 4, 6, 8, 12, 24, 72, 120, 168 hours postdose
Assessment of tic behaviors associated with TS using the Yale Global Tic Severity Scale (YGTSS) | Days 1, 7, 14, and 21

SECONDARY OUTCOMES:
Assessment of tic behaviors associated with TS using the Rush Video-based Tic Rating Scale (RTRS) | Days 1, 7, 14, and 21
Quantification of the premonitory urge phenomena associated with tics using the Premonitory Urge for Tics Scale (PUTS) | Days 1, 7, 14, and 21
Clinical Global Impression of Tourette Syndrome (CGI-TS) | Days 1, 7, 14, and 21
CogState computerized test to assess cognitive function | Day 1 at predose, 2.5 and 8 hours postdose; Day 14 at 8 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Principal Investigator — Neurocrine Biosciences
Locations (10):
- United States (10):
  - San Diego, California
  - Kissimmee, Florida
  - St. Petersburg, Florida
  - Naperville, Illinois
  - St Louis, Missouri
  - Lincoln, Nebraska
  - New York, New York
  - Rochester, New York
  - Petersburg, Virginia
  - Kirkland, Washington